CLINICAL TRIAL: NCT05086042
Title: Carpal Tunnel Syndrome in Patients With Psoriatic Arthritis; Ultrasonography and Magnetic Resonance Imaging Findings
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ezgi AKYILDIZ TEZCAN, M.D., Selcuk University
Other Study IDs: CTSINPSAUSMRI
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Carpal Tunnel Syndrome; Psoriatic Arthritis
Keywords: Carpal Tunnel Syndrome; Psoriatic Arthritis; Ultrasonography; magnetic resonance imaging
MeSH Terms: conditions — Carpal Tunnel Syndrome; Arthritis, Psoriatic | interventions — Ultrasonography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psoriatic arthritis patients
  Interventions: Diagnostic Test: Ultrasonography, Magnetic resonance imaging
- healthy volunteers
  Interventions: Diagnostic Test: Ultrasonography, Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Ultrasonography, Magnetic resonance imaging — The cross-sectional area of the median nerve was measured with US and MRI.

SUMMARY:
This study aimed to investigate relationship between CTS diagnosis with electrodiagnostic studies and median nerve's cross-sectional area measered by US and MRI in PsA patients.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a type of entrapment neuropathy, caused by compression of the median nerve in the carpal tunnel at the wrist1. It accounts for about 90% of all entrapment neuropathies. But there is no gold standard technique for diagnosing CTS. Electrodiagnostic studies (EDS) are generally used in differential diagnosis because the symptoms may be difficult to interpret. Unfortunetely EDS has some limitations. The factors can limit EDS are that it is not comfortable for patients and physicians, may require interventional procedures, need patient cooperation, provide limited information on the etiology of CTS, time consuming, and can not be used in some patient groups such as patients with dermatological contraindications. Recent years, magnetic resonance imaging (MRI) and ultrasonography (US) have facilitated the diagnosis of CTS. The median nerve cross-sectional area (CSA) measured by US or MRI has been found to be associated with CTS. However, there are studies with conflicting results regarding the median nerve CSA in patients with rheumatic diseases. Psoriatic arthritis (PsA), a kind of rheumatic disease, occurs in up to 30% of people with psoriasis and can have serious debilitating effects on the peripheral joints, spine, tendon insertions, and fingers. To our knowlage, any study didn't assess MRI measurements of median nerve CSA in PsA patients. In this study we aimed to assess CTS's US and MRI findings in patients with PsA and compare them healty controls.

ELIGIBILITY:
Inclusion Criteria:

* PsA patients according to the CASPAR criteria who consecutively applied to the FTR outpatient clinic for PsA follow-up and healthy volunteers who applied to the FTR outpatient clinic enrolled in the study.

Exclusion Criteria:

* Patients were excluded from the study if they had history of conditions associated with an increased incidence of CTS except PsA (diabetes mellitus, pregnancy, hypothyroidism, renal failure or other severe systemic diseases); history or clinical/electrophyscologic finding of radiculopathy, plexopathy, polyneuropathy or any nervous system diseases; history of fractures, severe trauma or surgical interventions involving the wrist; bifid median nerve on wrist imaging and under the age of 18, over the age of 65. There was no history of rheumatic disease in the healthy volunteer group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PsA patients according to the CASPAR criteria who consecutively applied to the FTR outpatient clinic for PsA follow-up and healthy volunteers who applied to the FTR outpatient clinic enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
The cross-sectional area of the median nerve measured by US and MRI | 12 months
  The measurement will be made at the pisiform bone level and with the continuous trace method.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Medicine, Konya, Turkey (Türkiye)